CLINICAL TRIAL: NCT01196026
Title: Immunogenicity and Safety Study of GSK Biologicals' Seasonal (2010-2011) Influenza Vaccine Fluarix™ in Children Previously Vaccinated With GSK Biologicals' H1N1 Vaccine Pandemrix™
Brief Title: Immunogenicity and Safety Study of Fluarix™ Vaccine in Children Who Have Previously Been Vaccinated With Pandemrix™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114451
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: Influenza; H1N1; Fluarix; Pandemrix
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (6):
- Fluarix 6-11 months Group (Experimental): Subjects previously vaccinated with Pandemrix vaccine, will receive one or two doses of Fluarix vaccine
  Interventions: Biological: Fluarix™
- Fluarix 12-35 months Group (Experimental): Subjects previously vaccinated with Pandemrix vaccine, will receive one or two doses of Fluarix vaccine
  Interventions: Biological: Fluarix™
- Fluarix 3-9 years Group (Experimental): Subjects previously vaccinated with Pandemrix vaccine, will receive one or two doses of Fluarix vaccine
  Interventions: Biological: Fluarix™
- Havrix Junior 6-11 months Group (Active Comparator): Subjects previously vaccinated with Pandemrix vaccine will receive two doses of Havrix Junior vaccine
  Interventions: Biological: Havrix™ Junior
- Havrix Junior 12-35 months Group (Active Comparator): Subjects previously vaccinated with Pandemrix vaccine will receive two doses of Havrix Junior vaccine
  Interventions: Biological: Havrix™ Junior
- Havrix Junior 3-9 years Group (Active Comparator): Subjects previously vaccinated with Pandemrix vaccine will receive two doses of Havrix Junior vaccine
  Interventions: Biological: Havrix™ Junior

INTERVENTIONS:
Biological: Fluarix™ — One or two intramuscular injections
  Arms: Fluarix 12-35 months Group; Fluarix 3-9 years Group; Fluarix 6-11 months Group
Biological: Havrix™ Junior — Two intramuscular injections
  Arms: Havrix Junior 12-35 months Group; Havrix Junior 3-9 years Group; Havrix Junior 6-11 months Group

SUMMARY:
This study is designed to assess the immunogenicity, reactogenicity and safety following vaccination with GSK Biologicals' Fluarix vaccine in children who have previously been vaccinated with two doses of Pandemrix at the age of 6 months-9 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having previously been immunized with two 0.25 mL doses of Pandemrix, given at least 21 days apart, at the age of 6 months to 9 years inclusive at the time of first vaccination.
* Subjects having received the last dose of Pandemrix at least six months prior to study enrolment.
* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the subjects.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Parent/LAR with access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.

Exclusion Criteria:

* Active participation in other clinical trials.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Planned administration of any vaccine 30 days prior and 30 days after any study vaccine administration.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to enrolment in this study or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned use during the study.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* History of seizures or progressive neurological disease.
* Subjects having received an H1N1v pandemic vaccine other than Pandemrix or having received the 2010/2011 seasonal influenza vaccine.
* Child in care.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2010-09-15; Primary Completion 2011-05-26 (Actual); Study Completion 2011-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- GSK Investigational Site, Rotterdam, Netherlands
- Sweden (6):
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Skellefteå
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Umeå

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Vesikari T, Richardus JH, Berglund J, Korhonen T, Flodmark CE, Lindstrand A, Silfverdal SA, Bambure V, Caplanusi A, Dieussaert I, Roy-Ghanta S, Vaughn DW. Immunogenicity and Safety of a Trivalent Inactivated Influenza Vaccine in Children 6 Months to 17 Years of Age, Previously Vaccinated with an AS03-Adjuvanted A(H1N1)Pdm09 Vaccine: Two Open-label, Randomized Trials. Pediatr Infect Dis J. 2015 Jul;34(7):774-82. doi: 10.1097/INF.0000000000000709. PMID 26069949
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114451 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114451 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114451 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114451 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114451 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114451 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primed subjects =subjects who had been previously vaccinated with a seasonal influenza vaccine whereas unprimed subjects had not.
  * children ≥ 9 years + primed children < 9 years=1 dose of Fluarix
  * unprimed children < 9 years=2 doses of Fluarix. To complete the vaccination schedule, a 2nd dose of Havrix vaccine was given outside the study setting
Pre-assignment Details: 162 subjects were enrolled in the study but only 154 subjects were vaccinated. The remaining 8 subjects gave their consent withdrawal and were not included in the study.Enrollment was stratified according to the age at first Pandemrix vaccination: 6-11 months, 12-35 months, 3-9 years. Also, subjects were grouped from 3-5 and from 6-9 years.
Groups:
- Fluarix 6-11 Months Group: Subjects aged 6 to 11 months and previously vaccinated with Pandemrix vaccine, will receive one or two doses of Fluarix™ vaccine depending on their priming status.
- Fluarix 12-35 Months Group: Subjects aged 12 to 35 months and previously vaccinated with Pandemrix vaccine, will receive one or two doses of Fluarix™ vaccine depending on their priming status.
- Fluarix 3-9 Years Group: Subjects aged 3 to 9 years and previously vaccinated with Pandemrix vaccine, will receive one or two doses of Fluarix™ vaccine depending on their priming status.
- Havrix Junior 6-11 Months Group: Subjects aged 6 to 11 months and previously vaccinated with Pandemrix vaccine will receive two doses of Havrix™ Junior vaccine.
- Havrix Junior 12-35 Months Group: Subjects aged 12 to 35 months and previously vaccinated with Pandemrix vaccine will receive two doses of Havrix™ Junior vaccine.
- Havrix Junior 3-9 Years Group: Subjects aged 3 to 9 years and previously vaccinated with Pandemrix vaccine will receive two doses of Havrix™ Junior vaccine.
Period: Overall Study
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Started | 10 | 44 | 23 | 10 | 43 | 24
Completed at Day 28 | 9 | 41 | 23 | 10 | 42 | 24
Completed | 9 | 36 | 23 | 10 | 42 | 24
Not Completed | 1 | 8 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Havrix Junior 6-11 Months Group: Subjects aged 12 to 35 months and previously vaccinated with Pandemrix vaccine will receive two doses of Havrix™ Junior vaccine.
- Havrix Junior 12-35 Months Group: Subjects aged 12-35 months and previously vaccinated with Pandemrix vaccine will receive two doses of Havrix Junior vaccine.
- Total: Total of all reporting groups
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Total
Number analyzed (Participants) | 10 | 44 | 23 | 10 | 43 | 24 | 154
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.0 (0.00) | 2.3 (0.52) | 6.4 (1.99) | 1.0 (0.00) | 2.4 (0.58) | 7.5 (1.53) | 3.58 (2.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 21 | 13 | 4 | 16 | 13 | 72
  Male | 5 | 23 | 10 | 6 | 27 | 11 | 82

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against H1N1 in All Subjects Receiving Fluarix Vaccine
Description: Antibody titers were expressed as Geometric mean titers (GMTs).
Time Frame: Day 0 and 28
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity at Day 28 which included all evaluable subjects for whom immunogenicity data at day 28 were available. The data presented here are only for the Fluarix All Ages Group. Similar data for other groups will be presented as Secondary Outcome Measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Fluarix All Ages Group: Subjects aged 6 months to 9 years and previously vaccinated with Pandemrix vaccine, will receive one or two doses of Fluarix vaccine depending on their priming status.
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 65
titer
  Day 0 |  |  |  |  |  |  | 120.7 [100.8 to 144.4]
  Day 28 |  |  |  |  |  |  | 1079.3 [915.8 to 1272.0]

2. Primary Outcome: Number of Subjects Seropositive for HI Antibodies Against H1N1 in All Subjects Receiving Fluarix Vaccine
Description: Seropositivity was defined as antibody titers greater than or equal to 1:10.
Time Frame: Day 0-28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 65
Participants
  Day 0 |  |  |  |  |  |  | 65
  Day 28 |  |  |  |  |  |  | 65

3. Primary Outcome: Number of Subjects Seroprotected for HI Antibodies Against H1N1 in All Subjects Receiving Fluarix Vaccine
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection.
Time Frame: Day 0-28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 65
Participants
  Day 0 |  |  |  |  |  |  | 63
  Day 28 |  |  |  |  |  |  | 65

4. Primary Outcome: Number of Subjects Seroconverted for HI Antibodies Against H1N1 in All Subjects Receiving Fluarix Vaccine
Description: A seroconverted subject was defined as a subject that had either a prevaccination (Day 0) titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 65
Participants |  |  |  |  |  |  | 55

5. Primary Outcome: Mean Geometric Increase (MGI) in HI Antibody Titers Against H1N1 in All Subjects Receiving Fluarix Vaccine
Description: MGI is defined as the geometric mean of the within-subject ratios of the post-vaccination (Day 28) reciprocal HI titer to the pre-vaccination (Day 0) reciprocal HI titer.
Time Frame: Day 28
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 65
ratio |  |  |  |  |  |  | 8.9 [7.1 to 11.2]

6. Secondary Outcome: HI Antibody Titers Against All Fluarix Vaccine Strains
Description: Antibody titers were expressed as GMTs. Vaccine strains included in the analysis were Flu A/CAL/7/09 H1N1 , FluB/Bri/60/08 Victoria, and Flu A/Vic/210/09 H3N2, further in this summary denoted as H1N1, Victoria and H3N2 strains, respectively.
Time Frame: Day 0 (for all groups) and Day 28 (for groups receiving Fluarix only)
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity at Day 28 which included all evaluable subjects for whom immunogenicity data at day 28 were available.
Measure: Mean (95% Confidence Interval); unit: titer
Groups:
- Havrix Junior All Ages Group: Subjects aged 6 months to 9 years and previously vaccinated with Pandemrix vaccine, will receive two doses of Havrix Junior vaccine.
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 7 | 35 | 23 | 10 | 43 | 24 | 65 | 77
titer
  H1N1 Day 0 | 176.6 [79.3 to 393.4] | 124.9 [97.1 to 160.5] | 102.0 [77.2 to 134.9] | 171.4 [118.9 to 247.2] | 186.5 [148.8 to 233.8] | 105.3 [75.4 to 147.0] | 120.7 [100.8 to 144.4] | 154.4 [129.8 to 183.7]
  H1N1 Day 28 | 1810.2 [775.2 to 4226.8] | 1345.0 [1141.9 to 1584.1] | 659.7 [524.1 to 830.3] | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6. | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6. | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6. | 1079.3 [915.8 to 1272.0] | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6.
  Victoria Day 0 | 16.4 [3.7 to 71.9] | 15.1 [10.6 to 21.5] | 21.9 [14.0 to 34.1] | 13.6 [7.6 to 24.6] | 19.1 [14.4 to 25.4] | 19.1 [12.3 to 29.6] | 17.4 [13.2 to 22.8] | 18.3 [14.8 to 22.7]
  Victoria Day 28 | 176.8 [28.1 to 1111.2] | 142.2 [93.5 to 216.2] | 188.8 [103.7 to 343.8] | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6. | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6. | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6. | 160.9 [115.0 to 225.2] | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6.
  H3N2 Day 0 | 5.0 [5.0 to 5.0] | 21.2 [13.7 to 32.8] | 31.0 [19.0 to 50.5] | 5.0 [5.0 to 5.0] | 8.9 [6.4 to 12.4] | 26.7 [16.6 to 42.9] | 20.8 [15.2 to 28.3] | 11.7 [8.9 to 15.2]
  H3N2 Day 28 | 88.4 [35.9 to 217.6] | 448.3 [265.9 to 755.8] | 518.6 [304.1 to 884.3] | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6. | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6. | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6. | 396.3 [276.3 to 568.5] | NA [NA to NA] — Data not planned to be collected at Day 28, but rather at Month 6.

7. Secondary Outcome: HI Antibody Titers Against H1N1 in Subjects Receiving Havrix Junior Vaccine
Description: Antibody titers were expressed as GMTs. Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains for subjects in groups receiving Fluarix vaccine and H1N1 strain for subjects in groups receiving Havrix Junior Vaccine.
Time Frame: Day 0 and Month 6
Population: Analysis was performed on According-to-Protocol (ATP) cohort for persistence at Month 6 which included all evaluable subjects for whom immunogenicity data at Month 6 were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
titer
  H1N1 Day 0 | 201.6 [81.1 to 501.1] | 126.4 [93.2 to 171.4] | 96.9 [73.9 to 126.9] | 172.8 [113.9 to 262.1] | 195.6 [155.1 to 246.6] | 100.3 [71.8 to 140.1] | 119.7 [97.9 to 146.3] | 154.6 [128.8 to 185.5]
  H1N1 Month 6 | 1437.0 [595.7 to 3466.6] | 565.5 [458.1 to 698.2] | 335.5 [253.1 to 444.7] | 93.4 [48.6 to 179.5] | 172.0 [127.9 to 231.4] | 74.3 [55.4 to 99.6] | 509.0 [416.9 to 621.5] | 120.7 [97.2 to 149.8]
  Victoria Day 0 | 17.8 [2.9 to 110.0] | 16.2 [10.6 to 24.6] | 21.6 [13.6 to 34.5] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 18.3 [13.5 to 24.8] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  Victoria Month 6 | 302.0 [115.6 to 788.8] | 148.4 [97.9 to 225.1] | 134.5 [82.2 to 220.1] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 154.1 [115.3 to 205.9] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Day 0 | 5.0 [5.0 to 5.0] | 20.3 [12.4 to 33.0] | 29.7 [17.9 to 49.2] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 20.3 [14.5 to 28.2] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Month 6 | 127.0 [70.1 to 230.0] | 160.0 [119.1 to 214.8] | 252.7 [186.3 to 342.8] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 186.8 [152.9 to 228.2] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.

8. Secondary Outcome: Number of Subjects Seropositive for HI Antibodies Against All Fluarix Vaccine Strains
Description: Seropositivity was defined as antibody titers greater than or equal to 1:10. Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains.
Time Frame: Day 0 (for all groups) and Day 28 (for groups receiving Fluarix only)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 7 | 35 | 23 | 10 | 43 | 24 | 65 | 77
Participants
  H1N1 Day 0 | 7 | 35 | 23 | 10 | 43 | 24 | 65 | 77
  H1N1 Day 28 | 7 | 35 | 23 | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | 65 | NA — Data not planned to be collected at Day 28, but rather at Month 6.
  Victoria Day 0 | 4 | 25 | 20 | 9 | 39 | 20 | 49 | 68
  Victoria Day 28 | 7 | 35 | 23 | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | 65 | NA — Data not planned to be collected at Day 28, but rather at Month 6.
  H3N2 Day 0 | 0 | 22 | 19 | 0 | 11 | 19 | 41 | 30
  H3N2 Day 28 | 7 | 35 | 23 | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | 65 | NA — Data not planned to be collected at Day 28, but rather at Month 6.

9. Secondary Outcome: Number of Subjects Seropositive for HI Antibodies Against H1N1 in Subjects Receiving Havrix Junior Vaccine
Description: Seropositivity was defined as antibody titers greater than or equal to 1:10. Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains for subjects in groups receiving Fluarix vaccine and H1N1 strain for subjects in groups receiving Havrix Junior Vaccine.
Time Frame: Day 0 and Month 6
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
Participants
  H1N1 Day 0 | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
  H1N1 Month 6 | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
  Victoria Day 0 | 3 | 21 | 19 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 43 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  Victoria Month 6 | 6 | 28 | 22 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 56 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Day 0 | 0 | 17 | 18 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 35 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Month 6 | 6 | 28 | 22 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 56 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.

10. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against All Fluarix Vaccine Strains in All Subjects Receiving Fluarix Vaccine
Description: A seroconverted subject was defined as a subject that had either a pre-vaccination (Day 0) titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer.
  Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains.
Time Frame: Day 28
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity at Day 28 which included all evaluable subjects for whom immunogenicity data at day 28 were available. Analysis was done only on those groups receiving the Fluarix vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 7 | 35 | 23 | 0 | 0 | 0 | 65 | 0
Participants
  H1N1 | 5 | 31 | 19 |  |  |  | 55 |
  Victoria | 7 | 30 | 18 |  |  |  | 55 |
  H3N2 | 7 | 35 | 22 |  |  |  | 64 |

11. Secondary Outcome: Number of Subjects Seroconverted for HI Antibodies Against H1N1 in Subjects Receiving Havrix Junior Vaccine
Description: A seroconverted subject was defined as a subject that had either a pre-vaccination (Day 0) titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer.
  Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains for subjects in groups receiving Fluarix vaccine and H1N1 strain for subjects in groups receiving Havrix Junior Vaccine.
Time Frame: Month 6
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
Participants
  H1N1 | 5 | 18 | 12 | 0 | 1 | 0 | 35 | 1
  Victoria | 5 | 22 | 15 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 42 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 | 6 | 22 | 18 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 46 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.

12. Secondary Outcome: Number of Subjects Seroprotected for HI Antibodies Against All Fluarix Vaccine Strains
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection. Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains.
Time Frame: Day 0 (for all groups) and Day 28 (for groups receiving Fluarix only)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 7 | 35 | 23 | 10 | 43 | 24 | 65 | 77
Participants
  H1N1 Day 0 | 7 | 33 | 23 | 10 | 43 | 24 | 63 | 77
  H1N1 Day 28 | 7 | 35 | 23 | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | 65 | NA — Data not planned to be collected at Day 28, but rather at Month 6.
  Victoria Day 0 | 2 | 5 | 7 | 1 | 9 | 7 | 14 | 17
  Victoria Day 28 | 7 | 35 | 21 | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | 63 | NA — Data not planned to be collected at Day 28, but rather at Month 6.
  H3N2 Day 0 | 0 | 17 | 13 | 0 | 6 | 12 | 30 | 18
  H3N2 Day 28 | 7 | 35 | 23 | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | NA — Data not planned to be collected at Day 28, but rather at Month 6. | 65 | NA — Data not planned to be collected at Day 28, but rather at Month 6.

13. Secondary Outcome: Number of Subjects Seroprotected for HI Antibodies Against H1N1 in Subjects Receiving Havrix Junior Vaccine
Description: A seroprotected subject was defined as a subject with a serum HI titer greater than or equal to 1:40 that usually is accepted as indicating protection. Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains for subjects in groups receiving Fluarix vaccine and H1N1 strain for subjects in groups receiving Havrix Junior Vaccine.
Time Frame: Day 0 and Month 6
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
Participants
  H1N1 Day 0 | 6 | 26 | 22 | 9 | 38 | 23 | 54 | 70
  H1N1 Month 6 | 6 | 28 | 22 | 8 | 36 | 21 | 56 | 65
  Victoria Day 0 | 2 | 5 | 7 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 14 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  Victoria Month 6 | 6 | 26 | 20 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 52 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Day 0 | 0 | 13 | 12 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 25 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Month 6 | 6 | 28 | 22 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 56 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.

14. Secondary Outcome: Mean Geometric Increase (MGI) in HI Antibody Titers Against All Fluarix Vaccine Strains in All Subjects Receiving Fluarix Vaccine
Description: MGI is defined as the geometric mean of the within-subject ratios of the post-vaccination (Day 28) reciprocal HI titer to the pre-vaccination (Day 0) reciprocal HI titer. Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains.
Time Frame: Day 28
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 7 | 35 | 23 | 0 | 0 | 0 | 65 | 0
ratio
  H1N1 | 10.2 [3.0 to 34.8] | 10.8 [7.9 to 14.7] | 6.5 [4.7 to 8.8] |  |  |  | 8.9 [7.1 to 11.2] |
  Victoria | 10.8 [5.9 to 19.6] | 9.4 [6.8 to 12.9] | 8.6 [5.5 to 13.6] |  |  |  | 9.3 [7.3 to 11.7] |
  H3N2 | 17.7 [7.2 to 43.5] | 21.1 [16.3 to 27.4] | 16.7 [11.4 to 24.6] |  |  |  | 19.1 [15.6 to 23.4] |

15. Secondary Outcome: Mean Geometric Increase (MGI) in HI Antibody Titers Against H1N1 in Subjects Receiving Havrix Junior Vaccine
Description: MGI is defined as the geometric mean of the within-subject ratios of the post-vaccination (Month 6) reciprocal HI titer to the pre-vaccination (Day 0) reciprocal HI titer.
  Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains for subjects in groups receiving Fluarix vaccine and H1N1 strain for subjects in groups receiving Havrix Junior Vaccine.
Time Frame: Month 6
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
ratio
  H1N1 | 7.1 [2.0 to 25.5] | 4.5 [3.3 to 6.0] | 3.5 [2.6 to 4.7] | 0.5 [0.4 to 0.8] | 0.9 [0.7 to 1.1] | 0.7 [0.7 to 0.8] | 4.3 [3.4 to 5.3] | 0.8 [0.7 to 0.9]
  Victoria | 17.0 [3.1 to 93.9] | 9.2 [5.9 to 14.2] | 6.2 [3.8 to 10.2] | NA [NA to NA] — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 8.4 [6.1 to 11.6] | NA [NA to NA] — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 | 25.4 [14.0 to 46.0] | 7.9 [5.5 to 11.4] | 8.5 [5.9 to 12.3] | NA [NA to NA] — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 9.2 [7.2 to 11.8] | NA [NA to NA] — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.

16. Secondary Outcome: Serum Neutralising Antibody Titers Against All Fluarix Vaccine Strains
Description: Antibody titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: Day 0 (for all groups) and Day 28 (for groups receiving Fluarix only)
Population: as for outcome 10
Measure: Geometric Mean (90% Confidence Interval); unit: titer
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 7 | 35 | 23 | 0 | 0 | 0 | 65 | 0
titer
  H1N1 Day 0: number analyzed (Participants) | 7 | 34 | 23 | 0 | 0 | 0 | 64 | 0
  H1N1 Day 0 | 359.1 [159.7 to 807.4] | 235.4 [180.5 to 307.0] | 237.6 [154.7 to 364.8] |  |  |  | 247.3 [199.6 to 306.5] |
  H1N1 Day 28: number analyzed (Participants) | 7 | 34 | 23 | 0 | 0 | 0 | 64 | 0
  H1N1 Day 28 | 5706.2 [3382.6 to 9626.0] | 5860.4 [5072.5 to 6770.7] | 2052.3 [1395.1 to 3019.0] |  |  |  | 4007.7 [3274.8 to 4904.6] |
  Victoria Day 0 | 20.2 [8.3 to 49.2] | 19.1 [13.9 to 26.2] | 25.4 [16.6 to 38.9] |  |  |  | 21.3 [16.8 to 26.9] |
  Victoria Day 28: number analyzed (Participants) | 7 | 34 | 23 | 0 | 0 | 0 | 64 | 0
  Victoria Day 28 | 49.3 [6.9 to 349.5] | 42.3 [20.9 to 85.5] | 80.8 [34.8 to 187.9] |  |  |  | 54.3 [33.0 to 89.3] |
  H3N2 Day 0 | 30.0 [13.5 to 66.9] | 84.9 [53.7 to 134.5] | 139.5 [100.8 to 193.0] |  |  |  | 90.5 [67.4 to 121.6] |
  H3N2 Day 28: number analyzed (Participants) | 7 | 34 | 23 | 0 | 0 | 0 | 64 | 0
  H3N2 Day 28 | 90.1 [50.1 to 162.0] | 1011.6 [509.5 to 2008.6] | 1229.9 [586.5 to 2579.3] |  |  |  | 832.9 [514.7 to 1347.8] |

17. Secondary Outcome: Serum Neutralising Antibody Titers Against H1N1 in Subjects Receiving Havrix Junior Vaccine
Description: Antibody titers were expressed as GMTs.] Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains for subjects in groups receiving Fluarix vaccine and H1N1 strain for subjects in groups receiving Havrix Junior Vaccine.
Time Frame: Day 0 and Month 6
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
titer
  H1N1 Day 0: number analyzed (Participants) | 6 | 27 | 22 | 9 | 38 | 23 | 55 | 70
  H1N1 Day 0 | 419.1 [172.0 to 1021.2] | 254.8 [184.0 to 352.8] | 221.2 [145.0 to 337.6] | 292.0 [170.8 to 499.1] | 441.3 [317.5 to 613.5] | 212.8 [142.3 to 318.1] | 254.2 [200.2 to 322.9] | 329.3 [260.0 to 417.2]
  H1N1 Month 6 | 5080.1 [2169.7 to 11894.4] | 2359.7 [1852.0 to 3006.4] | 892.2 [585.7 to 1359.0] | 292.6 [173.6 to 493.0] | 528.9 [377.5 to 741.0] | 221.6 [155.0 to 316.8] | 1748.2 [1347.3 to 2268.4] | 368.3 [290.1 to 467.5]
  Victoria Day 0 | 21.4 [7.2 to 64.0] | 20.7 [13.9 to 30.7] | 26.1 [16.8 to 40.6] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 22.7 [17.4 to 29.7] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  Victoria Month 6 | 284.5 [89.4 to 905.6] | 140.0 [81.7 to 240.0] | 113.1 [58.2 to 219.7] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 138.9 [95.2 to 202.6] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Day 0 | 34.1 [13.6 to 85.3] | 78.4 [47.0 to 131.1] | 136.5 [97.4 to 191.3] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 89.2 [65.5 to 121.5] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Month 6 | 264.1 [136.0 to 512.9] | 618.2 [435.1 to 878.5] | 638.2 [381.1 to 1068.8] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 571.5 [435.5 to 749.8] | NA [NA to NA] — Titers were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.

18. Secondary Outcome: Number of Subjects Seropositive for Serum Neutralising Antibodies Against All Fluarix Vaccine Strains
Description: Seropositivity was defined as antibody titers greater than or equal to 1:28.
Time Frame: Day 0 (for all groups) and Day 28 (for groups receiving Fluarix only)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 7 | 35 | 23 | 0 | 0 | 0 | 65 | 0
Participants
  H1N1 Day 0: number analyzed (Participants) | 7 | 34 | 23 | 0 | 0 | 0 | 64 | 0
  H1N1 Day 0 | 7 | 34 | 23 |  |  |  | 64 |
  H1N1 Day 28: number analyzed (Participants) | 7 | 34 | 23 | 0 | 0 | 0 | 64 | 0
  H1N1 Day 28 | 7 | 34 | 23 |  |  |  | 64 |
  Victoria Day 0 | 1 | 5 | 7 |  |  |  | 13 |
  Victoria Day 28: number analyzed (Participants) | 7 | 34 | 23 | 0 | 0 | 0 | 64 | 0
  Victoria Day 28 | 3 | 15 | 12 |  |  |  | 30 |
  H3N2 Day 0 | 4 | 26 | 22 |  |  |  | 52 |
  H3N2 Day28: number analyzed (Participants) | 7 | 34 | 23 | 0 | 0 | 0 | 64 | 0
  H3N2 Day28 | 7 | 34 | 23 |  |  |  | 64 |

19. Secondary Outcome: Number of Subjects Seropositive for Serum Neutralising Antibodies Against H1N1 in Subjects Receiving Havrix Junior Vaccine
Description: Seropositivity was defined as antibody titers greater than or equal to 1:28. Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains for subjects in groups receiving Fluarix vaccine and H1N1 strain for subjects in groups receiving Havrix Junior Vaccine.
Time Frame: Day 0 and Month 6
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
Participants
  H1N1 Day 0: number analyzed (Participants) | 6 | 27 | 22 | 9 | 38 | 23 | 55 | 70
  H1N1 Day 0 | 6 | 27 | 22 | 9 | 38 | 23 | 55 | 70
  H1N1 Month 6 | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
  Victoria Day 0 | 1 | 5 | 7 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 13 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  Victoria Month 6 | 6 | 28 | 18 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 52 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Day 0 | 4 | 20 | 21 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 45 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 Month 6 | 6 | 28 | 22 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 56 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.

20. Secondary Outcome: Number of Subjects Seroconverted for Serum Neutralising Antibodies Against All Fluarix Vaccine Strains in Subjects Receiving Fluarix
Description: Seroconverted subject was a subject with a minimum 4-fold increase in titer at post-vaccination for neutralizing antibody response.
Time Frame: Day 28
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 7 | 34 | 23 | 0 | 0 | 0 | 64 | 0
Participants
  H1N1: number analyzed (Participants) | 7 | 33 | 23 | 0 | 0 | 0 | 63 | 0
  H1N1 | 6 | 33 | 17 |  |  |  | 56 |
  Victoria | 3 | 11 | 11 |  |  |  | 25 |
  H3N2 | 4 | 32 | 16 |  |  |  | 52 |

21. Secondary Outcome: Number of Subjects Seroconverted for Serum Neutralising Antibodies Against H1N1 in Subjects Receiving Havrix Junior Vaccine
Description: Seroconverted subject was a subject with a minimum 4-fold increase in titer at post-vaccination for neutralizing antibody response.
  Vaccine strains included in the analysis were H1N1, Victoria and H3N2 strains for subjects in groups receiving Fluarix vaccine and H1N1 strain for subjects in groups receiving Havrix Junior Vaccine.
Time Frame: Month 6
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group | Fluarix All Ages Group | Havrix Junior All Ages Group
Number analyzed (Participants) | 6 | 28 | 22 | 9 | 38 | 23 | 56 | 70
Participants
  H1N1: number analyzed (Participants) | 6 | 27 | 22 | 9 | 38 | 23 | 55 | 70
  H1N1 | 5 | 22 | 10 | 0 | 2 | 0 | 37 | 2
  Victoria | 6 | 23 | 13 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 42 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.
  H3N2 | 5 | 21 | 13 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine. | 39 | NA — Results were available only against H1N1 antigen in subjects receiving Havrix Junior Vaccine.

22. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed include: pain, redness and swelling. Any is any symptom regardless of intensity. Grade 3 was defined as a symptom that prevented normal activity.above 50 millimeter.
Time Frame: During the 7 days (Day 0 - 6) after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, on subjects that had completed their symptom sheet for the respective vaccine dose only.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 10 | 43 | 23 | 10 | 43 | 24
Participants
  Any Pain | 3 | 28 | 21 | 5 | 19 | 14
  Grade 3 Pain | 0 | 1 | 1 | 0 | 1 | 0
  Any Redness | 7 | 33 | 19 | 2 | 15 | 9
  Grade 3 Redness | 2 | 8 | 6 | 0 | 0 | 0
  Any Swelling | 5 | 23 | 11 | 1 | 10 | 5
  Grade 3 Swelling | 1 | 3 | 2 | 0 | 0 | 0

23. Secondary Outcome: Duration of Any Solicited Local Symptom
Description: Duration was expressed as median number of days the symptom persisted. Solicited local symptoms assessed include: pain, redness and swelling.
Time Frame: During the 7 days (Days 0 - 6) after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, on subjects that had completed their symptom sheet and reported the respective symptom only.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 6 | 30 | 20 | 5 | 19 | 14
days
  Pain [Dose 1]: number analyzed (Participants) | 3 | 23 | 20 | 5 | 19 | 14
  Pain [Dose 1] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 4.0]
  Redness [Dose 1]: number analyzed (Participants) | 6 | 30 | 16 | 2 | 15 | 9
  Redness [Dose 1] | 4.0 [1.0 to 6.0] | 3.0 [1.0 to 7.0] | 3.0 [1.0 to 6.0] | 1.5 [1.0 to 2.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 5.0]
  Swelling [Dose 1]: number analyzed (Participants) | 5 | 18 | 9 | 1 | 10 | 5
  Swelling [Dose 1] | 2.0 [1.0 to 5.0] | 3.0 [1.0 to 6.0] | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 3.0]
  Pain [Dose 2]: number analyzed (Participants) | 2 | 21 | 14 | 5 | 19 | 14
  Pain [Dose 2] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — None of the subjects from the Havrix Groups received a second vaccine dose within the frame of this study. | NA [NA to NA] — None of the subjects from the Havrix Groups received a second vaccine dose within the frame of this study. | NA [NA to NA] — None of the subjects from the Havrix Groups received a second vaccine dose within the frame of this study.
  Redness [Dose 2]: number analyzed (Participants) | 4 | 23 | 13 | 5 | 19 | 14
  Redness [Dose 2] | 3.0 [3.0 to 7.0] | 3.0 [1.0 to 6.0] | 2.0 [1.0 to 5.0] | NA [NA to NA] — None of the subjects from the Havrix Groups received a second vaccine dose within the frame of this study. | NA [NA to NA] — None of the subjects from the Havrix Groups received a second vaccine dose within the frame of this study. | NA [NA to NA] — None of the subjects from the Havrix Groups received a second vaccine dose within the frame of this study.
  Swelling [Dose 2]: number analyzed (Participants) | 2 | 16 | 8 | 5 | 19 | 14
  Swelling [Dose 2] | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 4.0] | NA [NA to NA] — None of the subjects from the Havrix Groups received a second vaccine dose within the frame of this study. | NA [NA to NA] — None of the subjects from the Havrix Groups received a second vaccine dose within the frame of this study. | NA [NA to NA] — None of the subjects from the Havrix Groups received a second vaccine dose within the frame of this study.

24. Secondary Outcome: Number of Subjects Less Than 6 Years Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed include diarrhoea, drowsiness, irritability, loss of appetite and fever. Any was defined as any symptom regardless of intensity; any fever was axillary temperature greater than or equal to 37.5 degrees celsius. Grade 3 was a symptom preventing normal everyday activity; grade 3 loss of appetite was not eating at all; grade 3 fever was axillary temperature above 39 degrees celsius. Related was any symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7 days (Days 0-6) after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, on subjects aged less than 6 years that had completed their symptom sheet for the respective vaccine dose only.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 10 | 43 | 11 | 10 | 43 | 2
Participants
  Any Diarrhoea | 5 | 8 | 2 | 2 | 7 | 0
  Grade 3 Diarrhoea | 0 | 0 | 0 | 0 | 1 | 0
  Related Diarrhoea | 5 | 3 | 1 | 2 | 3 | 0
  Any Drowsiness | 6 | 16 | 2 | 2 | 15 | 0
  Grade 3 Drowsiness | 0 | 3 | 1 | 0 | 2 | 0
  Related Drowsiness | 5 | 10 | 2 | 2 | 9 | 0
  Any Irritability | 6 | 20 | 4 | 5 | 14 | 0
  Grade 3 Irritability | 0 | 1 | 0 | 0 | 2 | 0
  Related Irritability | 5 | 14 | 3 | 4 | 10 | 0
  Any Loss of Appetite | 6 | 14 | 4 | 3 | 6 | 0
  Grade 3 Loss of Appetite | 0 | 1 | 0 | 0 | 0 | 0
  Related Loss of Appetite | 4 | 8 | 4 | 2 | 3 | 0
  Any Fever | 5 | 14 | 4 | 3 | 11 | 0
  Grade 3 Fever | 1 | 1 | 1 | 0 | 0 | 0
  Related Fever | 4 | 11 | 3 | 0 | 4 | 0

25. Secondary Outcome: Duration of Any Solicited General Symptom Experienced by Subjects Less Than 6 Years Old
Description: Duration was expressed as median number of days the symptom persisted. Solicited general symptoms assessed include diarrhoea, drowsiness, irritability, loss of appetite and fever.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: as for outcome 24
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 5 | 14 | 3 | 5 | 15 | 0
days
  Diarrhoea [Dose 1]: number analyzed (Participants) | 3 | 6 | 1 | 2 | 7 | 0
  Diarrhoea [Dose 1] | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0] | 3.5 [1.0 to 6.0] | 1.0 [1.0 to 3.0] |
  Drowsiness [Dose 1]: number analyzed (Participants) | 4 | 11 | 1 | 2 | 15 | 0
  Drowsiness [Dose 1] | 1.5 [1.0 to 6.0] | 1.0 [1.0 to 4.0] | 3.0 [3.0 to 3.0] | 2.0 [2.0 to 2.0] | 2.0 [1.0 to 6.0] |
  Irritability [Dose 1]: number analyzed (Participants) | 4 | 14 | 3 | 5 | 14 | 0
  Irritability [Dose 1] | 2.5 [1.0 to 4.0] | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 5.0] |
  Loss of Appetite [Dose 1]: number analyzed (Participants) | 5 | 11 | 3 | 3 | 6 | 0
  Loss of Appetite [Dose 1] | 2.0 [1.0 to 6.0] | 3.0 [1.0 to 5.0] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 7.0] | 1.5 [1.0 to 3.0] |
  Fever [Dose 1]: number analyzed (Participants) | 3 | 10 | 2 | 3 | 11 | 0
  Fever [Dose 1] | 4.0 [1.0 to 6.0] | 1.5 [1.0 to 3.0] | 1.5 [1.0 to 2.0] | 2.0 [2.0 to 2.0] | 2.0 [1.0 to 6.0] |
  Diarrhoea [Dose 2]: number analyzed (Participants) | 4 | 4 | 1 | 5 | 15 | 0
  Diarrhoea [Dose 2] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0] | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. |
  Drowsiness [Dose 2]: number analyzed (Participants) | 4 | 9 | 2 | 5 | 15 | 0
  Drowsiness [Dose 2] | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. |
  Irritability [Dose 2]: number analyzed (Participants) | 5 | 12 | 2 | 5 | 15 | 0
  Irritability [Dose 2] | 2.0 [2.0 to 7.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. |
  Loss of Appetite [Dose 2]: number analyzed (Participants) | 4 | 9 | 2 | 5 | 15 | 0
  Loss of Appetite [Dose 2] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0] | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. |
  Fever [Dose 2]: number analyzed (Participants) | 3 | 9 | 2 | 5 | 15 | 0
  Fever [Dose 2] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 7.0] | 1.0 [1.0 to 1.0] | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. | NA [NA to NA] — None of the subjects in any of the Havrix Groups received a second vaccine dose. |

26. Secondary Outcome: Number of Subjects Above 6 Years Reported Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed include arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering, sweating and fever. Any was defined as any symptom regardless of intensity; any fever was axillary temperature greater than or equal to 37.5 degrees celsius. Grade 3 was a symptom preventing normal everyday activity; grade 3 fever was axillary temperature above 39 degrees celsius. Related was any symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, on subjects aged above 6 years that had completed their symptom sheet for the respective vaccine dose only.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 0 | 0 | 12 | 0 | 0 | 22
Participants
  Any Arthralgia |  |  | 0 |  |  | 0
  Grade 3 Arthralgia |  |  | 0 |  |  | 0
  Related Arthralgia |  |  | 0 |  |  | 0
  Any Fatigue |  |  | 5 |  |  | 8
  Grade 3 Fatigue |  |  | 0 |  |  | 0
  Related Fatigue |  |  | 4 |  |  | 6
  Any Gatrointestinal Symptoms |  |  | 1 |  |  | 1
  Grade 3 Gatrointestinal Symptoms |  |  | 0 |  |  | 0
  Related Gatrointestinal Symptoms |  |  | 1 |  |  | 1
  Any Headache |  |  | 4 |  |  | 4
  Grade 3 Headache |  |  | 0 |  |  | 0
  Related Headache |  |  | 3 |  |  | 3
  Any Myalgia |  |  | 1 |  |  | 2
  Grade 3 Myalgia |  |  | 0 |  |  | 0
  Related Myalgia |  |  | 1 |  |  | 2
  Any Shivering |  |  | 2 |  |  | 0
  Grade 3 Shivering |  |  | 0 |  |  | 0
  Related Shivering |  |  | 2 |  |  | 0
  Any Sweating |  |  | 0 |  |  | 0
  Grade 3 Sweating |  |  | 0 |  |  | 0
  Related Sweating |  |  | 0 |  |  | 0
  Any Fever |  |  | 3 |  |  | 0
  Grade 3 Fever |  |  | 0 |  |  | 0
  Related Fever |  |  | 2 |  |  | 0

27. Secondary Outcome: Duration of Any Solicited General Symptom Experienced by Subjects Above 6 Years Old
Description: Duration was expressed as median number of days the symptom persisted. Solicited general symptoms assessed include fatigue, gastrointestinal symptoms, headache, myalgia, shivering and fever.
Time Frame: During a 7-day follow-up period (Day 0-6) after vaccination
Population: as for outcome 26
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 8
days
  Fatigue [Dose 1] |  |  | 1.5 [1.0 to 5.0] |  |  | 1.0 [1.0 to 2.0]
  Fatigue [Dose 2]: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 8
  Fatigue [Dose 2] |  |  | 4.0 [1.0 to 7.0] |  |  | NA [NA to NA] — Dose 2 involved subjects in Group receiving Fluarix vaccine.
  Gastrointestinal Symptoms [Dose 1]: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  Gastrointestinal Symptoms [Dose 1] |  |  | 2.0 [2.0 to 2.0] |  |  | 1.0 [1.0 to 1.0]
  Gastrointestinal symptoms [Dose 2] |  |  | NA [NA to NA] — None of the subjects aged above 6 years in this group experienced this symptom |  |  | NA [NA to NA] — Dose 2 involved subjects in Group receiving Fluarix vaccine.
  Headache [Dose 1]: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 4
  Headache [Dose 1] |  |  | 3.0 [2.0 to 4.0] |  |  | 3.0 [1.0 to 7.0]
  Headache [Dose 2]: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 8
  Headache [Dose 2] |  |  | 3.5 [3.0 to 4.0] |  |  | NA [NA to NA] — Dose 2 involved subjects in Group receiving Fluarix vaccine.
  Myalgia [Dose 1]: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 2
  Myalgia [Dose 1] |  |  | NA [NA to NA] — None of the subjects aged above 6 years in this group experienced this symptom. |  |  | 1.0 [1.0 to 1.0]
  Myalgia [Dose 2]: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 8
  Myalgia [Dose 2] |  |  | 1.0 [1.0 to 1.0] |  |  | NA [NA to NA] — Dose 2 involved subjects in Group receiving Fluarix vaccine.
  Shivering [Dose 1]: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 8
  Shivering [Dose 1] |  |  | 1.0 [1.0 to 1.0] |  |  | NA [NA to NA] — None of the subjects aged above 6 years in this group experienced this symptom.
  Shivering [Dose 2] |  |  | NA [NA to NA] — None of the subjects aged above 6 years in this group experienced this symptom |  |  | NA [NA to NA] — Dose 2 involved subjects in Group receiving Fluarix vaccine.
  Fever [Dose 1] |  |  | 1.0 [1.0 to 1.0] |  |  | NA [NA to NA] — None of the subjects aged above 6 years in this group experienced this symptom.
  Fever [Dose2]: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 8
  Fever [Dose2] |  |  | 1.0 [1.0 to 1.0] |  |  | NA [NA to NA] — Dose 2 involved subjects in Group receiving Fluarix vaccine.

28. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Any was defined as any symptom regardless of intensity or relationship to vaccination. Grade 3 was a symptom preventing normal everyday activity. Related was any symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 28 day follow-up period (Day 0-27) after vaccination
Population: The analysis was performed on the Total Vaccinated Cohort which included all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 10 | 44 | 23 | 10 | 43 | 24
Participants
  Any AEs | 6 | 20 | 7 | 3 | 15 | 7
  Grade 3 AEs | 3 | 4 | 1 | 0 | 1 | 1
  Related AEs | 2 | 1 | 2 | 0 | 1 | 0

29. Secondary Outcome: Number of Subjects Reporting Medically-Attended Events (MAEs), Adverse Events of Specific Interest (AESIs)/ Potential Immune Mediated Diseases (pIMDs) and Adverse Events (AEs) of Special Interest
Description: MAEs: subject received medical attention defined as hospitalisation, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason.
  AESIs/pIMD: includes both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Adverse events of special interest include both convulsion and anaphylaxis.
Time Frame: During the entire study period (up to Month 6)
Population: The analysis was performed on the Total Vaccinated Cohort which included all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 10 | 44 | 23 | 10 | 43 | 24
Participants
  MAEs | 4 | 11 | 2 | 3 | 7 | 1
  AESIs / pIMDs | 0 | 0 | 0 | 0 | 0 | 0
  AEs of special interest | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs: medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Up to Day 28
Population: The analysis was performed on the Total Vaccinated Cohort which included all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 10 | 44 | 23 | 10 | 43 | 24
Participants | 0 | 1 | 0 | 0 | 0 | 0

31. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: as for outcome 30
Time Frame: Up to Month 6
Population: The analysis was performed on the Total Vaccinated Cohort which included all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Number analyzed (Participants) | 10 | 44 | 23 | 10 | 43 | 24
Participants | 1 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed throughout the study period (from the beginning of the study up to Month 6). Systematically and non-systematically assessed frequent adverse events (AEs) were assessed during 7 days and 28 days post-vaccination.
Description: The following systematically assessed non-serious AEs were assessed only in subjects aged less than 6 years old: diarrhoea, drowsiness, irritability and loss of appetite. The following systematically assessed non-serious AEs were assessed only in subjects aged above 6 years old: fatigue, gastrointestinal symptoms, headache, myalgia and shivering.
Arm/Group | Fluarix 6-11 Months Group | Fluarix 12-35 Months Group | Fluarix 3-9 Years Group | Havrix Junior 6-11 Months Group | Havrix Junior 12-35 Months Group | Havrix Junior 3-9 Years Group
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/44 | 0/23 | 0/10 | 0/43 | 0/24
Other Adverse Events (participants affected / at risk) | 10/10 | 41/44 | 23/23 | 9/10 | 34/43 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix 6-11 Months Group (N=10) | Fluarix 12-35 Months Group (N=44) | Fluarix 3-9 Years Group (N=23) | Havrix Junior 6-11 Months Group (N=10) | Havrix Junior 12-35 Months Group (N=43) | Havrix Junior 3-9 Years Group (N=24)
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fluarix 6-11 Months Group (N=10) | Fluarix 12-35 Months Group (N=44) | Fluarix 3-9 Years Group (N=23) | Havrix Junior 6-11 Months Group (N=10) | Havrix Junior 12-35 Months Group (N=43) | Havrix Junior 3-9 Years Group (N=24)
Pain (General disorders) | 3 | 28/43 | 21 | 5 | 19 | 14
Redness (General disorders) | 7 | 33/43 | 19 | 2 | 15 | 9
Swelling (General disorders) | 5 | 23/43 | 11 | 1 | 10 | 5
Diarrhoea (General disorders) | 5 | 8/43 | 2/11 | 2 | 7 | 0/2
Drowsiness (General disorders) | 6 | 16/43 | 2/11 | 2 | 15 | 0/2
Irritability (General disorders) | 6 | 20/43 | 4/11 | 5 | 14 | 0/2
Loss of Appetite (General disorders) | 6 | 14/43 | 4/11 | 3 | 6 | 0/2
Fever (General disorders) | 5 | 14/43 | 4/11 | 3 | 11 | 0/2 — For subjects less than 6 years old
Upper respiratory tract infection (Infections and infestations) | 2 | 9 | 0 | 0 | 6 | 0
Gastroenteritis (Infections and infestations) | 0 | 4 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lip haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tooth discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Varicella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.